CLINICAL TRIAL: NCT03542331
Title: Histological and Transcriptional Changes Caused by Endometrial Flushing With Lipiodol: A Cross Over Study
Brief Title: Endometrial Effects of Lipiodol
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017.lipiodol.flush
Record Dates: First submitted 2018-04-13; First posted 2018-05-31 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Female Infertility
MeSH Terms: conditions — Infertility, Female | interventions — Ethiodized Oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Other): The control group wille have a mock catheter introduction between day 6 and 8 of the cycle without any Lipiodol flush
  Interventions: Device: Mock catheter
- Intervention group (Experimental): The intervention group will undergo endometrial flushing with Lipiodol between day 6 and 8 of the cycle
  Interventions: Drug: Lipiodol

INTERVENTIONS:
Drug: Lipiodol — Endometrial flushing with Lipiodol between day 6 and 8 of the cycle
  Arms: Intervention group
Device: Mock catheter — Introduction of a mock catheter in the uterus between day 6 and 8 of the cycle
  Arms: Control group

SUMMARY:
The goal is to investigate whether endometrial flushing with Lipiodol enhances fertility. Therefore, anatomo-pathological, histochemical and transcriptional changes of the endometrium after Lipiodol bathing in a general population of healthy volunteers will be determined.

DETAILED DESCRIPTION:
A single-centre, cross-over, open-label trial will be performed. Healthy volunteers, fulfilling the inclusion/exclusion criteria, will be asked to do blood samples and ultrasounds for the detection of the LH (luteinizing hormone) surge in a natural cycle. The intervention group will undergo endometrial flushing with Lipiodol between day 6 and 8 of the cycle, while the control group between day 6 and 8 of the cycle will have a mock catheter introduction without any Lipiodol flush. An endometrial biopsy will be performed 7 days after the LH peak in all the participants. Furthermore, all the participants will undergo one cycle with flushing and one cycle with introduction of a mock catheter but without flushing with any medication. The wash-out period between the 2 biopsies will be 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Women aged ≥18 and <36 years
* Regular cycle (25-35 days)
* Signed informed consent
* Participants can be included only once in the trial
* Contraceptive: barrier method only.

Exclusion Criteria:

* known iodine allergy
* Body mass index 30 or ≤18.5
* Smoking
* Previous diagnosis of PCO (Polycystic Ovary Syndrome) (>12 antral follicles in one ovary, Rotterdam criteria 2003)
* Previous diagnosis of endometriosis, uterine malformations or intrauterine pathologies (submucosal fibroids, endometrial polyps, and intrauterine adhesions)
* Systemic diseases such as thyroid dysfunction
* Breast-feeding or pregnancy within the last 6 months
* Intrauterine devices (IUD)
* History of recurrent miscarriage
* Known history of infertility
* Previous uterine surgery
* Pregnancy wish during the course of the study
* Women who have been previously enrolled in the trial
* Those unable to comprehend the investigational nature of the proposed study

Ages: 18 Years to 36 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Anatomo-pathological changes of the endometrium after Lipiodol bathing | 7 days after LH peak
  To determine whether the treatment with lipiodol alters the leukocyte population. Changes in the uterine dendritic cell population, collections of macrophages and an increased number of inflammatory cells will be investigated. A sub-ephitelial re-location of lymphocytes (CD3-CD7 and CD8 (CD: Cluster of Differentiation)) will be looked for.
Histochemical changes of the endometrium after Lipiodol bathing | 7 days after LH peak
  The immunohistochemistry for the key implantation factors, the subsequent molecular markers will be examined: estrogen receptors (ER) (α/β), progesterone receptors (PR) (A, B), prolactine (PRL), insulin-like growth factor binding protein-1 (IGF-BP1), leukaemia inhibitory factor (LIF), Mucins (MUC1), integrin αVβ3, vascular endothelial growth factor (VEG-F), transforming growth factor (TGF-β1).
Transcriptional changes of the endometrium after Lipiodol bathing | 7 days after LH peak
  RNA sequencing

CONTACTS AND LOCATIONS:
Locations (1):
- Universitair Ziekenhuis Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided